CLINICAL TRIAL: NCT00300027
Title: A Phase I Study to Determine the Safety, Pharmacokinetics and Pharmacodynamics of BMS-582664 in Combination With 5-Fluorouracil/Leucovorin and Irinotecan or Oxaliplatin for Patients With Advanced or Metastatic Cancer
Brief Title: Study of BMS-582664 in Combination With Either FOLFIRI or FOLFOX for Gastrointestinal (GI) Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA182-007
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2007-09

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Advanced Gastrointestinal Malignancies
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — brivanib

INTERVENTIONS:
Drug: BMS-582664

SUMMARY:
The purpose of this study is to define the recommended dose of BMS-582664 that could be safely combined with 5-fluorouracil, leucovorin, and irinotecan (FOLFIRI) or 5-fluorouracil, leucovorin, and oxaliplatin (FOLFOX) chemotherapy regimens in patients with advanced gastrointestinal malignancies and to evaluate the safety profile, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of these combinations.

ELIGIBILITY:
Inclusion Criteria:

* Good performance status
* Advanced colorectal, pancreatic, esophageal or gastric cancer
* Tissue for analyses
* Adequate bone marrow, hepatic, renal function
* 4-6 weeks since prior therapy
* Adequate protection for women of child bearing potential (WOCBP)

Exclusion Criteria:

* Brain metastasis
* Thromboembolic disease
* Cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-04; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety (vitals, labs, physical examination [PE], electrocardiogram [ECG]) every week (qw)
Echocardiogram every 2 cycles (q 2 cycles)

SECONDARY OUTCOMES:
Tumor response (q 2 cycles)
PK parameters (during 1st cycle)
PD markers (weekly)
Fluorodeoxyglucose positron emission tomography (FDG-PET) (3 scans prior to C3)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Los Angeles, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Iowa City, Iowa
  - Local Institution, Durham, North Carolina
  - Local Institution, Temple, Texas